CLINICAL TRIAL: NCT04957797
Title: Anatomic and Biomechanical Investigation on Anterior Cruciate Ligament: A Cadaveric Study
Brief Title: Anatomic and Biomechanical Investigation on ACL: A Cadaveric Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2019056
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Nine matched-paired fresh frozen human cadaveric knees were randomly distributed into two groups: Flat-tunnel (FLT) group and round-tunnel (ROT) group. One knee from each pair was reamed with flat tunnel, while the contralateral knee was reamed with round tunnel.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROT-Group (Other): reamed with round tunnel
  Interventions: Procedure: round tunnel
- FLT-Group (Experimental): reamed with flat tunnel
  Interventions: Procedure: flat tunnel

INTERVENTIONS:
Procedure: round tunnel — reamed with round tunnel
  Arms: ROT-Group
Procedure: flat tunnel — reamed with flat tunnel
  Arms: FLT-Group

SUMMARY:
The present study was aimed to investigate the kinematics differences between round-tunnel (ROT) and flat-tunnel (FLT) techniques and compare the influence to the anterior root of lateral meniscus (ARLM ) in anterior cruciate ligament (ACL) reconstruction when using hamstring graft.

DETAILED DESCRIPTION:
Nine matched pairs of fresh-frozen cadaveric knees were evaluated for the kinematics of intact, ACL-sectioned, and either ROT or FLT reconstructed knees. The graft bundles for FLT technique were separately tensioned. A 6 degrees of freedom robotic system was used to assess knee laxity: (1) 134-N anterior tibial load at 0°, 15°, 30°, 60°, and 90°of knee ﬂexion. (2) 10-Nm of valgus torque followed by 5-Nm of internal rotation torque simulates a pivot-shift test at 15°, 30°. (3) 5-Nm internal and external rotation torques at 0°, 15°, 30°, 60°, and 90°. (4) 10-Nm varus and valgus torques at 15°, 30°. Coverage of ACL tibial footprint and areas of ARLM attachment before and after reaming were measured using three-dimensional isotropic MRI scanning.

ELIGIBILITY:
Inclusion Criteria:

* intact knee with no previous injures

Exclusion Criteria:

* those with ligamentous injury or a limited range of motion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
simulated pivot-shift test | within 1 hour after surgery
  10-Nm of valgus torque followed by 5-Nm of internal rotation torque simulates a pivot-shift test at 15°, 30° of knee ﬂexion
simulated KT-2000 arthrometer | within 1 hour after surgery
  134-N anterior tibial load simulates a KT-2000 arthrometer at 0°, 15°, 30°, 60°, and 90°of knee ﬂexion
internal and external rotation | within 1 hour after surgery
  5-Nm internal and external rotation torques at 0°, 15°, 30°, 60°, and 90° of knee ﬂexion
varus and valgus | within 1 hour after surgery
  10-Nm varus and valgus torques at 15°, 30°of knee ﬂexion
average percentage of ACL tibial footprint coverage | within 1 hour after surgery
  Coverage of ACL tibial footprint and areas of ARLM attachment before and after reaming were measured using three-dimensional isotropic MRI scanning post-operation

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided